CLINICAL TRIAL: NCT00793819
Title: A Double-Blind, Placebo-Controlled Phase 2 Study of Silodosin 8 mg Daily for the Treatment of Nocturia in Men With Benign Prostatic Hyperplasia
Brief Title: A Study of Silodosin 8 mg Daily for the Treatment of Nocturia in Men With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SI08005
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-02

CONDITIONS: Nocturia; Prostatic Hyperplasia
Keywords: nocturia; BPH; benign prostate hyperplasia; nocturia in men with benign prostate hyperplasia
MeSH Terms: conditions — Nocturia; Prostatic Hyperplasia | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Silodosin (Experimental)
  Interventions: Drug: silodosin
- 2 Placebo (Placebo Comparator)
  Interventions: Drug: silodosin

INTERVENTIONS:
Drug: silodosin — α1-adrenergic antagonist
  Other Names: Rapaflo

SUMMARY:
Silodosin is compared to placebo to determine if it is safe and effective for the treatment of nighttime urination (nocturia) in men with BPH

DETAILED DESCRIPTION:
This will be a multi-center, double-blind, placebo controlled, parallel, 12 week treatment trial in men with signs and symptoms of benign prostatic hyperplasia and nocturia. The following procedures are utilized; physical exams, electrocardiograms, clinical laboratory tests, vital signs, urinary diary, Pittsburgh Quality of Sleep Index, Nocturia Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Males in good general health and at least 50 years of age, with symptoms of moderate to severe BPH and nocturia (>=2 episodes per night)

Exclusion Criteria:

* Medical conditions that would confound the efficacy evaluation.
* Medical conditions in which it would be unsafe to use an alpha-blocker.
* The use of concomitant drugs that would confound the efficacy evaluation.
* The use of concomitant drugs that would be unsafe with this alpha-blocker.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Caramelli, MS, Study Director — Watson Pharmaceuticals
Locations (27):
- United States (27):
  - Watson Investigational Site, Huntsville, Alabama
  - Watson Investigational Site, Laguna Hills, California
  - Watson Investigational Site, San Diego, California
  - Watson Investigational Site, Aventura, Florida
  - Watson Investigational Site, Clearwater, Florida
  - Watson Investigational Site, Orlando, Florida
  - Watson Investigational Site, Marietta, Georgia
  - Watson Investigational Site, Sandy Springs, Georgia
  - Watson Investigational Site, Coeur d'Alene, Idaho
  - Watson Investigational Site, West Des Moines, Iowa
  - Watson Investigational Site, Paducah, Kentucky
  - Watson Investigational Site, Greenbelt, Maryland
  - Watson Investigational Site, Troy, Michigan
  - Watson Investigational Site, Missoula, Montana
  - Watson Investigational Site, Omaha, Nebraska
  - Watson Investigational Site, Las Vegas, Nevada
  - Watson Investigational Site, Lawrenceville, New Jersey
  - Watson Investigational Site, Albuquerque, New Mexico
  - Watson Investigational Site, Bay Shore, New York
  - Watson Investigational Site, New York, New York
  - Watson Investigational Site, Williamsville, New York
  - Watson Investigational Site, Concord, North Carolina
  - Watson Investigational Site, Salisbury, North Carolina
  - Watson Investigational Site, Bethany, Oklahoma
  - Watson Investigational Site, Bala-Cynwyd, Pennsylvania
  - Watson Investigational Site, Myrtle Beach, South Carolina
  - Watson Investigational Site, Burien, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Silodosin 8mg: Silodosin 8mg daily
- Placebo: 1 placebo capsule daily
Period: Overall Study
Arm/Group | Silodosin 8mg | Placebo
Started | 111 | 98
Completed | 97 | 89
Not Completed | 14 | 9
Not completed — Adverse Event | 8 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silodosin 8mg | Placebo | Total
Number analyzed (Participants) | 111 | 98 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 62 | 125
  >=65 years | 48 | 36 | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.03) | 64.2 (8.92) | 64.4 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 111 | 98 | 209
Region of Enrollment [Number; unit: participants]
  United States | 111 | 98 | 209

OUTCOME MEASURES:

1. Primary Outcome: Change in Nocturia Episodes
Time Frame: 12 weeks
Population: The number of participants for analysis is determined by Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Silodosin 8mg | Placebo
Number analyzed (Participants) | 112 | 97
episodes | -1.2 (1.35) | -1.0 (1.44)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Silodosin 8mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/111 | 1/98
Other Adverse Events (participants affected / at risk) | 39/111 | 21/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silodosin 8mg (N=111) | Placebo (N=98)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Multiple Bone Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silodosin 8mg (N=111) | Placebo (N=98)
Retrograde Ejaculation (Reproductive system and breast disorders) | 24 (24) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 4 (5) | 3 (4)
Fatigue (General disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5)
Urinary Track Infection (Infections and infestations) | 0 (0) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Upper Respiratory Track Infection (Infections and infestations) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less